CLINICAL TRIAL: NCT06215326
Title: Short-term Effects of Preoperative Exercise in Moderate-to-high Perioperative Risk Lung Cancer Patients(PRE-EXELUCA): a Multicenter Prospective Randomized Controlled Clinical Trial
Brief Title: Short-term Effects of Preoperative Exercise in Moderate-to-high Perioperative Risk Lung Cancer Patients
Acronym: PRE-EXELUCA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY2023-535
Record Dates: First submitted 2023-12-20; First posted 2024-01-22 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2023-12

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; preoperative exercise; moderate-to-high perioperative risk; cardiorespiratory function; postoperative outcomes
MeSH Terms: conditions — Lung Neoplasms | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the study intervention, this study was an open trial and was not blinded to the patients and study executives. Only the outcome assessors and statistical analysts of the study will be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Moderate-intensity Continuous Training (MICT) Group (Experimental): MICT plan is containing usual care protocol and additional complete a total of 12 supervised moderate-intensity continuous training sessions in 2-3 weeks.
  Interventions: Behavioral: moderate-intensity continuous training
- High-intensity Interval Training (HIIT) Group (Experimental): HIIT plan is containing usual care protocol and additional complete a total of 12 supervised high-intensity interval training training sessions in 2-3 weeks.
  Interventions: Behavioral: high-intensity interval training
- Usual care group (No Intervention): Usual care is including smoking cessation instruction, respiratory exercise, review by a specialist nurse, meeting with the surgeon and anesthetist, and receiving information about preparing for surgery.

INTERVENTIONS:
Behavioral: moderate-intensity continuous training — Participants in MICT group will need to additional complete a total of 12 supervised training sessions in 2-3 weeks.After a warm-up of 5 minutes at 50% at peak WR, the patient start exercising at 60%-70% peak WR for 30-40 minutes (four 5-8 minutes sets, with a 2-min rest in between), and then the patients cooled down for 5 minutes at 50% peak WR. Moderate-intensity exercise training intensity control at 55-74% HRmax or 40-69% VO2peak or PRE12-13 as recommended by guidelines.
  Other Names: MICT
  Arms: Moderate-intensity Continuous Training (MICT) Group
Behavioral: high-intensity interval training — Participants in HIIT group will need to additional complete a total of 12 supervised training sessions in 2-3 weeks.After a 5-minute warm-up at 50% at peak WR, the patients complete 20 series of vigorous-intensity sprint (80%-100% peak WR for 30-60s) separated by a low-intensity recovery (30% peak WR or completely rest for 15s), and then the patients cooled down for 5 minutes at 50% peak WR. Participants will begin training at a relatively moderate intensity (60%-65% peak WR) for the first 3 sessions and gradually increase to the target intensity beginning on the 4th session. Intensity control of high-intensity exercise training at 75-90% HRmax or 70-85% VO2peak or PRE14-16 as recommended by guidelines.
  Other Names: HIIT
  Arms: High-intensity Interval Training (HIIT) Group

SUMMARY:
The goal of this clinical trail is to compare the effects of preoperative exercise training of different intensities on short-term cardiorespiratory function and postoperative outcomes in patients scheduled for lung resections.

DETAILED DESCRIPTION:
Guangdong Provincial People's Hospital will be the lead center, with an additional 3 hospitals designated as satellite centers for the study. To sum up, these centers will recruit a total of 100 consenting patients. Following informed consent and baseline testing, participants will be randomized into one of the three groups in a 2:1:1 ratio: MICT, HIIT, or usual care (UC).

Participants in the MICT and HIIT groups perform a total of 12 sessions of supervised exercise training, while participants randomized to the UC group receive no extra rehabilitation or physical activity. All participants are followed-up at the completion of the intervention period.Primary outcomes including cardiopulmonary exercise function and pulmonary function will be measured at diagnosis (lung cancer patients scheduled for surgical treatment) (V1), baseline (V2), and post-intervention (V3). The baseline assessment includes medical history and examination. To lessen the psychological burden of the study on the patients, the baseline examination phase could not be repeated if the examinations had been completed during the screening phase and the date of completion was within 7 days prior to enrollment. The patient's postoperative complications, chest tube removal time and hospital length of stay (LOS) will be recorded on the day of discharge (V4). Patient-reported outcomes (PROs) will be measured at baseline (V2), post-intervention (V3), day of discharge (V4), 1 month postoperative (V5), and 3 months postoperative (V6) with ongoing follow-up. Participant blood samples and diaphragm ultrasound will be retained at baseline(V2) and post-intervention (V3) as available. Postoperative deaths will be followed up by telephone on the day of discharge (V4), 3 months postoperatively (V6), 1 year postoperatively (V7), 3 years postoperatively (V8), and 5 years postoperatively (V9).

ELIGIBILITY:
Inclusion Criteria:

1. Age>18 years.
2. Suspected or confirmed primary lung cancer with scheduled surgical treatment.
3. Moderate-to-high perioperative risk, defined as FEV1<60% of predicted value (wedge) or ppo FEV1<60% of predicted value (lobectomy/segmentectomy) or VO2peak<20 ml/kg/ min.
4. Sign informed consent and accept to comply with the requirements of the study protocol.
5. Completion of a baseline Complete cardiopulmonary exercise testing (CPET).

Exclusion Criteria:

1. Concurrent or previous history of other malignant tumors.
2. Life expectancy less than 1 year.
3. Dementia; infirmity; or inability to participate in sports (musculoskeletal limitations, namely, injuries, frailty, and weakness).
4. Inability to maintain exercise training.
5. Irregular vital signs (heart rate: < 40 or > 120 bpm at rest; blood pressure: systolic blood pressure > 200 mm Hg or diastolic pressure > 110 mm Hg; T: ≥ 38.5 or ≤ 36◦C; SpO2 ≤ 90%).
6. Currently enrolling in any other clinical trials.
7. Patient refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
cardiopulmonary fitness | baseline，2 weeks
  The post-training change in cardiorespiratory fitness will be measured by the VO2peak in ml/kg/min.VO2peak will be evaluated by a cardiopulmonary exercise test.
pulmonary function | baseline，2 weeks
  Pulmonary function will be measured as the first step of the CPET. Predicted postoperative (PPO) lung functions will be calculated by the Forced Expiratory Volume in one second (FEV1). Pulmonary function in patients scheduled for wedge resection will be assessed as a predicted percentage of FEV1. Whereas participants planning to have segmentectomy or lobectomy will be evaluated with PPO FEV1 as a percentage of predicted value.

SECONDARY OUTCOMES:
postoperative complications | 1 week postoperative
  Postoperative complications will be recorded and graded specifically according to a modified version of the Thoracic Mortality and Morbidity (TMM) classification system, and related treatments will be recorded, with statistics on the incidence of TMM grade 2 or higher complications. In addition, chest tube duration and hospital LOS will be recorded.
postoperative mortality | 3 months, 1 year, 3 years and 5 years postoperative
  Postoperative mortality will be recorded by calling.
patient-reported outcomes | baseline，2 weeks, 1 week postoperative, 1 month postoperative and 3 months postoperative
  The MD Anderson Symptom Inventory-Lung Cancer (MDASI-LC), a validated lung cancer-specific scale, will be utilized to assesses patients' symptoms to measure patient-reported outcomes(PROs).MDASI-LC includes 16 symptom items with scores ranging from 0 (no symptom) to 10 (worst symptom imaginable) and six functional items with scores ranging from 0 (no interference) to 10 (complete interference).

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Drevet G, Belaroussi Y, Duruisseaux M, Chalabreysse L, Grima R, Maury JM, Tronc F. Futile lobectomies following video-thoracoscopic exploration for indeterminate pulmonary nodules: a retrospective study. J Thorac Dis. 2022 Aug;14(8):2826-2834. doi: 10.21037/jtd-21-1789. PMID 36071782
- [Result] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Result] Xia C, Dong X, Li H, Cao M, Sun D, He S, Yang F, Yan X, Zhang S, Li N, Chen W. Cancer statistics in China and United States, 2022: profiles, trends, and determinants. Chin Med J (Engl). 2022 Feb 9;135(5):584-590. doi: 10.1097/CM9.0000000000002108. PMID 35143424
- [Result] Howington JA, Blum MG, Chang AC, Balekian AA, Murthy SC. Treatment of stage I and II non-small cell lung cancer: Diagnosis and management of lung cancer, 3rd ed: American College of Chest Physicians evidence-based clinical practice guidelines. Chest. 2013 May;143(5 Suppl):e278S-e313S. doi: 10.1378/chest.12-2359. PMID 23649443
- [Result] Brunelli A, Refai MA, Salati M, Sabbatini A, Morgan-Hughes NJ, Rocco G. Carbon monoxide lung diffusion capacity improves risk stratification in patients without airflow limitation: evidence for systematic measurement before lung resection. Eur J Cardiothorac Surg. 2006 Apr;29(4):567-70. doi: 10.1016/j.ejcts.2006.01.014. Epub 2006 Feb 14. PMID 16481190
- [Result] Brunelli A, Charloux A, Bolliger CT, Rocco G, Sculier JP, Varela G, Licker M, Ferguson MK, Faivre-Finn C, Huber RM, Clini EM, Win T, De Ruysscher D, Goldman L; European Respiratory Society and European Society of Thoracic Surgeons joint task force on fitness for radical therapy. ERS/ESTS clinical guidelines on fitness for radical therapy in lung cancer patients (surgery and chemo-radiotherapy). Eur Respir J. 2009 Jul;34(1):17-41. doi: 10.1183/09031936.00184308. PMID 19567600
- [Result] Berry MF, Villamizar-Ortiz NR, Tong BC, Burfeind WR Jr, Harpole DH, D'Amico TA, Onaitis MW. Pulmonary function tests do not predict pulmonary complications after thoracoscopic lobectomy. Ann Thorac Surg. 2010 Apr;89(4):1044-51; discussion 1051-2. doi: 10.1016/j.athoracsur.2009.12.065. PMID 20338305
- [Result] Licker M, Schnyder JM, Frey JG, Diaper J, Cartier V, Inan C, Robert J, Bridevaux PO, Tschopp JM. Impact of aerobic exercise capacity and procedure-related factors in lung cancer surgery. Eur Respir J. 2011 May;37(5):1189-98. doi: 10.1183/09031936.00069910. Epub 2010 Sep 16. PMID 20847073
- [Result] Brunelli A, Kim AW, Berger KI, Addrizzo-Harris DJ. Physiologic evaluation of the patient with lung cancer being considered for resectional surgery: Diagnosis and management of lung cancer, 3rd ed: American College of Chest Physicians evidence-based clinical practice guidelines. Chest. 2013 May;143(5 Suppl):e166S-e190S. doi: 10.1378/chest.12-2395. PMID 23649437
- [Result] Odor PM, Bampoe S, Gilhooly D, Creagh-Brown B, Moonesinghe SR. Perioperative interventions for prevention of postoperative pulmonary complications: systematic review and meta-analysis. BMJ. 2020 Mar 11;368:m540. doi: 10.1136/bmj.m540. PMID 32161042
- [Result] Liu Z, Qiu T, Pei L, Zhang Y, Xu L, Cui Y, Liang N, Li S, Chen W, Huang Y. Two-Week Multimodal Prehabilitation Program Improves Perioperative Functional Capability in Patients Undergoing Thoracoscopic Lobectomy for Lung Cancer: A Randomized Controlled Trial. Anesth Analg. 2020 Sep;131(3):840-849. doi: 10.1213/ANE.0000000000004342. PMID 31348053
- [Result] Licker M, Karenovics W, Diaper J, Fresard I, Triponez F, Ellenberger C, Schorer R, Kayser B, Bridevaux PO. Short-Term Preoperative High-Intensity Interval Training in Patients Awaiting Lung Cancer Surgery: A Randomized Controlled Trial. J Thorac Oncol. 2017 Feb;12(2):323-333. doi: 10.1016/j.jtho.2016.09.125. Epub 2016 Oct 19. PMID 27771425
- [Result] Steffens D, Beckenkamp PR, Hancock M, Solomon M, Young J. Preoperative exercise halves the postoperative complication rate in patients with lung cancer: a systematic review of the effect of exercise on complications, length of stay and quality of life in patients with cancer. Br J Sports Med. 2018 Mar;52(5):344. doi: 10.1136/bjsports-2017-098032. Epub 2018 Feb 1. PMID 29437041
- [Result] Gravier FE, Smondack P, Prieur G, Medrinal C, Combret Y, Muir JF, Baste JM, Cuvelier A, Boujibar F, Bonnevie T. Effects of exercise training in people with non-small cell lung cancer before lung resection: a systematic review and meta-analysis. Thorax. 2022 May;77(5):486-496. doi: 10.1136/thoraxjnl-2021-217242. Epub 2021 Aug 24. PMID 34429375
- [Result] Granger C, Cavalheri V. Preoperative exercise training for people with non-small cell lung cancer. Cochrane Database Syst Rev. 2022 Sep 28;9(9):CD012020. doi: 10.1002/14651858.CD012020.pub3. PMID 36170564
- [Result] Ligibel JA, Bohlke K, May AM, Clinton SK, Demark-Wahnefried W, Gilchrist SC, Irwin ML, Late M, Mansfield S, Marshall TF, Meyerhardt JA, Thomson CA, Wood WA, Alfano CM. Exercise, Diet, and Weight Management During Cancer Treatment: ASCO Guideline. J Clin Oncol. 2022 Aug 1;40(22):2491-2507. doi: 10.1200/JCO.22.00687. Epub 2022 May 16. PMID 35576506
- [Result] Cavalheri V, Granger CL. Exercise training as part of lung cancer therapy. Respirology. 2020 Nov;25 Suppl 2:80-87. doi: 10.1111/resp.13869. Epub 2020 Jun 1. PMID 32567236
- [Result] Mendoza TR, Wang XS, Lu C, Palos GR, Liao Z, Mobley GM, Kapoor S, Cleeland CS. Measuring the symptom burden of lung cancer: the validity and utility of the lung cancer module of the M. D. Anderson Symptom Inventory. Oncologist. 2011;16(2):217-27. doi: 10.1634/theoncologist.2010-0193. Epub 2011 Feb 1. PMID 21285393